CLINICAL TRIAL: NCT03413540
Title: Dose-Dependent Effects of Jumping on Bone Health in Premenopausal Women
Brief Title: Effects of Jumping on Bone Health in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, San Marcos (Other)
Responsible Party: Principal Investigator, Kara Witzke, Professor, Kinesiology, California State University, San Marcos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1SC3GM084705 (NIH)
Record Dates: First submitted 2018-01-21; First posted 2018-01-29 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Osteoporosis, Osteopenia
Keywords: jumping; bone health
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — acj6 protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Group 1 (Experimental): 10-cm step, 10 reps
  Interventions: Other: Jump
- Group 2 (Experimental): 10-cm step, 50 reps
  Interventions: Other: Jump
- Group 3 (Experimental): 10-cm step, 100 reps
  Interventions: Other: Jump
- Group 4 (Experimental): 20-cm step, 10 reps
  Interventions: Other: Jump
- Group 5 (Experimental): 20-cm step, 50 reps
  Interventions: Other: Jump
- Group 6 (Experimental): 20-cm step, 100 reps
  Interventions: Other: Jump
- Group 7 (Experimental): 30-cm step, 10 reps
  Interventions: Other: Jump
- Group 8 (Experimental): 30-cm step, 50 reps
  Interventions: Other: Jump
- Group 9 (Experimental): 30-cm step, 100 reps
  Interventions: Other: Jump
- Group 10 (No Intervention): Control

INTERVENTIONS:
Other: Jump — Drop jump from step
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6; Group 7; Group 8; Group 9

SUMMARY:
This study evaluates the longitudinal, dose-dependent effects of jumping on bone health in young women. The women will be divided into 9 groups of varying jump height and repetitions, with a tenth group serving as control.

DETAILED DESCRIPTION:
Over 1 million hip and spine fractures each year are associated with osteoporosis, a disease of low bone mass that contributes to increased morbidity, mortality and economic strain on our medical system. Effective low-cost prevention strategies such as bone-loading exercise, could lower the incidence of osteoporotic fractures without an increase in medical costs, and provide an alternative to drug therapy. Activity associated with high magnitude forces such as fast running and jumping, have been shown to increase hip bone mass by 1.2%-4% in premenopausal women which may translate into a 20-30% reduction in hip fracture risk. In addition, high impact exercise may also produce benefits that are maintained long-term. However, a specific exercise prescription for improving bone health has not been determined.

To date, no single study has examined the interactive effects of jump magnitude (height) and jump number (repetitions) on bone mineral density by systematically varying the height and number of jumps performed. In addition, no study has evaluated the effects of loading exercise on multiple measures of bone health, in order to quantify the effects of exercise on bone strength, apart from bone mineral density. Determining the optimal dose of jump exercise for improving bone strength will allow the investigators to determine a specific exercise prescription for bone health in premenopausal women and will be useful in future projects that intend to employ jump training to target bone health. The long-term objective of this line of research is to determine how impact loading improves bone quality to ultimately reduce fracture risk.

This study is a randomized, controlled, trial to compare the effects of a 9-month supervised exercise program using three levels of load magnitude (4", 8", 12" jump height) and three load repetitions (10, 50, 100 jumps per session), on three dimensions of bone health (bone density, remodeling and strength) in 300 premenopausal women aged 18-42y. Bone density is the most widely recognized dimension of bone health and clinically accepted index of fracture risk. Bone remodeling reflects the dynamic state of bone and can predict fracture risk independent of bone density. Bone strength, represented by Femur Strength Index, is a reflection of the geometry and structural competence of bone.

Low-cost osteoporosis prevention strategies including jumping exercises, could lower the incidence of osteoporotic fractures without an increase in medical costs, and provide an alternative to drug therapy. This project will allow the investigators to determine the minimum effective dose of jumping exercise required to benefit bone health in premenopausal women and will lead to future research on how exercise improves bone quality and reduces fracture risk.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal with a history of regular menses (10-12 cycles/year)

Exclusion Criteria:

* Current smoking
* Obesity (BMI > 30 kg/m2) or underweight (BMI < 18 kg/m2)
* Use of medications known to affect bone metabolism including thyroid hormone, thiazide diuretics, aromatase inhibitors, hormone replacement therapy, selective estrogen receptor modulators (SERMS) and bisphosphonates within the previous 6 months. (Note: Women currently using hormonal birth control (e.g. estrogen, progesterone, depot medroxyprogesterone acetate) for at least the previous 12 months will not be excluded from participation, but will be asked to continue with their current method throughout the study period).
* Chronic disorders that affect bone metabolism and/or the ability to participate in exercise training such as diabetes, hyperparathyroidism, uncontrolled hypothyroidism, balance difficulties, use of narcotic medication.
* Regular participation in exercise associated with a large volume of jumping (i.e., volleyball, basketball, high-impact aerobics, plyometrics, gymnastics, etc) within the past year.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pre-menopausal women
Enrollment: 357 (Actual)
Dates: Start 2008-09-28 (Actual); Primary Completion 2012-06-13 (Actual); Study Completion 2012-06-13 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Change from baseline bone mineral density at 9 months
  Bone mineral density using dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Bone remodeling | Change from baseline bone formation and resorption markers at 9 months
  Bone formation and resorption markers in blood
Bone strength | Change from baseline femur strength index at 9 months
  Femur strength Index (FSI) calculated from DXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Kara A Witzke, PhD, Principal Investigator — Oregon State University - Cascades

IPD SHARING:
Plan to Share IPD: Undecided